CLINICAL TRIAL: NCT04153084
Title: Comparative Study of Effectiveness and Safety of Different Endoscopic Preparations Used in Pediatric Colonoscopy
Brief Title: Study of Different Endoscopic Preparations Used in Pediatric Colonoscopy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fundación Pública Andaluza para la gestión de la Investigación en Sevilla (Other)
Responsible Party: Sponsor
Other Study IDs: FIS-POL-2017-01
Record Dates: First submitted 2019-11-04; First posted 2019-11-06 (Actual); Last update posted 2019-11-08 (Actual); Status verified 2019-09

CONDITIONS: Digestive Illness
Keywords: Pediatric colonoscopy; Endoscopic preparations; PEG; Sodium picosulfate; Bohm solution; Movicol; Picoprep; Colonoscopic examination
MeSH Terms: interventions — polyethylene glycol 4000; Electrolytes; polyethylene glycol 3350; picosulfate sodium

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- High volume electrolytes Polyethylene Glycol (PEG 4000) cohort: Pediatric patients who have prepared for a colonoscopy during the years 2018-2019 using high volume electrolytes PEG (Bohm solution®) endoscopic preparation, as part of a diagnostic procedure not related to this study.
  Interventions: Drug: Polyethylene Glycol 4000 with electrolytes
- Low volume electrolytes PEG (PEG 3350) cohort: Pediatric patients who have prepared for a colonoscopy during the years 2018-2019 using low volume electrolytes PEG (Movicol®) endoscopic preparation, as part of a diagnostic procedure not related to this study.
  Interventions: Drug: PEG-3350 with electrolytes
- Sodium picosulfate cohort: Pediatric patients who have prepared for a colonoscopy during the years 2018-2019 using sodium picosulfate (Picoprep®) endoscopic preparation, as part of a diagnostic procedure not related to this study.
  Interventions: Drug: Sodium picosulfate

INTERVENTIONS:
Drug: Polyethylene Glycol 4000 with electrolytes — The high volume electrolytes PEG will be administered at a 4 mg/kg dose the day before the procedure in 4-8 hours.
  Other Names: Bohm solution®
  Groups: High volume electrolytes Polyethylene Glycol (PEG 4000) cohort
Drug: PEG-3350 with electrolytes — The low volume electrolytes PEG will be administered at a 4 mg/kg dose the day before the procedure in 4-8 hours.
  Other Names: Movicol®
  Groups: Low volume electrolytes PEG (PEG 3350) cohort
Drug: Sodium picosulfate — The Sodium picosulfate will be administered the day before the procedure at different doses depending on the patient´s age:
  * From 1 to 2 years old: ¼ sachet reconstituted in ¼ glass of water/juice in the afternoon (15:00 h) and ¼ sachet reconstituted in ¼ glass of water/juice 6 hours later (21:00 h)
  * From 2 to 4 years old: ½ sachet in ½ glass of water/juice in the afternoon and ½ sachet in ½ glass of water/juice at night.
  * From 4 to 9 years old: 1 sachet in 1 glass of water/juice in the afternoon and ½ sachet in ½ glass of water/juice at night.
  * Of 9 years old and older: 1 sachet in the afternoon and 1 sachet at night.
  Other Names: Picoprep®
  Groups: Sodium picosulfate cohort

SUMMARY:
The aim of this study is to evaluate the quality, acceptance, tolerability and adverse effects of colonoscopy preparations with the different available preparation guidelines.

ELIGIBILITY:
Inclusion Criteria:

* From 1 to 16 years old.
* Patients that signed the informed consent form.

Exclusion Criteria:

* Urgent colonoscopy
* History of intestinal resection
* Nephropathy, heart disease or metabolic syndrome.

Ages: 1 Year to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric patients who have undergone a colonoscopic exploration during the years 2018-2019, as part of a diagnostic process not related to the study.
Sampling Method: Probability Sample
Enrollment: 126 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-12-15 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluate the quality of the colonoscopy preparations in our autonomic community comparing different preparation guidelines : Boston Scale | From November 2018 to December 2019
  The quality of the preparations will be measured using the Boston Bowel Preparation Scale (BBPS), semiquantitative evaluation of the cleanliness of the three colon sections (left, transverse, right) using a score from 0 to 3, giving a total score of 0 (without preparation) to 9 (optimal) and it´s done by two independent observers.

SECONDARY OUTCOMES:
Evaluate the acceptance of the different preparations. | From November 2018 to December 2019
  The acceptance will be measured using a questionnaire and a quantity record, the questonnaire is made by three items: flavour, odour and volume while the quantity record measures the quantity of preparation ingested by the participant.
Evaluate the tolerance of the different preparations. | From November 2018 to December 2019
  The tolerance will be measured using a questionnaire and a symptoms record, with a score from 0 (terrible tolerance) to 3 (good tolerance) for each of its items, that are the following: abdominal pain, nausea and vomit, intestinal noises, abdominal distension, burps, flatulences, urgent bowel movements and tenesmus.
Evaluate the security of the different preparations. | From November 2018 to December 2019
  The security will be measured analysing the existence of adverse effects due to the different preparations.

CONTACTS AND LOCATIONS:
Overall Officials: Alejandro Rodríguez Martínez, Principal Investigator — Hospital Universitario Virgen Rocío
Locations (8):
- Spain (8):
  - Hospital Universitario Puerta del Mar, Cadiz, Cádiz
  - Complejo Hospitalario Torrecárdenas, Almería
  - Hospital Materno-Infantil de Badajoz, Badajoz
  - Hospital Universitario Reina Sofía, Córdoba
  - Hospital Universitario Virgen de las Nieves, Granada
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Universitario Virgen del Rocío, Seville
  - Instituto Hispalense de Pediatría, Seville